CLINICAL TRIAL: NCT00894127
Title: Sputum Labeling Utilizing Synthetic Meso Tetra (4-Carboxyphenyl) Porphine (TCPP) for Detection of Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomoda Inc. (Industry)
Collaborators: Alquest (Industry); Quintiles, Inc. (Industry); Radiology Associates of Albuquerque (Other); New Mexico Technical Institute of Mining and Technology (Unknown); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MODA-001
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Porphyrin; Fluorescence; Diagnostic; Sputum Cytology; Early Detection
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyPath Assay of Deep-Lung Sputum Sample (Experimental): Deep-lung sputum was obtained from two cohorts, including (1) high-risk control group comprised of individuals not diagnosed but at high risk for lung cancer (n=102) and, (2) cancer group comprised of individuals with confirmed lung cancer diagnosis (n=26), was labeled in exact manner with TCPP and evaluated to detect red fluorescent [ie, cancer] cells (RFCs) from deep-lung sputum samples.
  Interventions: Device: CyPath

INTERVENTIONS:
Device: CyPath — CyPath diagnostic assay for the early detection of lung cancer using sputum

SUMMARY:
Primary Objective:

* To determine the clinical sensitivity and specificity of the Biomoda CyPath™ Early Lung Cancer Detection Assay using sputum specimens from two cohorts of participants and estimate the required sample size to finalize a protocol for a pivotal study.

Secondary Objectives:

* To assess the capability of the Biomoda CyPath™ Early Lung Cancer Detection Assay in a clinical setting to identify cancer cells, as assessed by TCPP labeled cancer cells demonstrating red fluorescence under a microscope with ultraviolet (UV) light being observed with a FITC (Fluorescein isothiocyanate) Filter.
* To assess the capability of the Biomoda CyPath™ Early Lung Cancer Detection Assay to detect pre-invasive cancer in comparison with PAP sputum cytology and routine CT scan.

DETAILED DESCRIPTION:
Meso Tetra (4-Carboxyphenyl) Porphine (TCPP) is a porphyrin that can label cancer cells by reacting to the increased number of low-density lipoproteins coating the surface of cancer cells and the porous nature of the cancer cell membrane, causing the cell to fluoresce under specific wavelengths of light. The primary objective of this clinical trial was to determine the clinical sensitivity and specificity of the CyPath® Lung Cancer Detection Assay ("CyPath® Assay") using sputum specimens from two cohorts of Participants. The Study design included a protocol to assess the capability of the Biomoda CyPath® Lung Cancer Detection Assay to detect cancer in comparison with routine high-resolution, low-dose Computed Tomography (LDCT) scans.

Optimization of the Assay can lead to improved sensitivity and specificity. Increase in sample size and evaluation of the entire sputum sample can increase data collection and differentiation between cohorts. Technicians in the current Study examined 12 slides containing approximately 600,000 cells. The average sputum sample pellet translates to a potential of approximately 3.5 million cells for evaluation. Evaluating the full sputum sample with the CyPath® Assay can be accomplished through flow cytometry and would increase the capture and analysis of exfoliated cancer cells in the sample. In-house studies evaluated samples from five different cancer cell lines using flow cytometry. Preliminary results showed that cancer cell lines were detected with significant fluorescence apart from normal cell fluorescence. Refinements for using the flow cytometer include optimizing the liquid-based assay and sample analysis and focus on concentration, incubation time and optimal sample volume.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veterans
* Study Participants must be willing to provide primary care physician contact information and agree to have medical information released if indicated
* Meet requirements of one of the two cohorts in the study:
* Cohort 1: Heavy Smoker

  * Defined as 20 pack years or greater (e.g., 1 pack/day for 20 years or 2 packs/day for 10 years).
* Cohort 2: Known Lung Cancer

  * Recently diagnosed with Stage I - IV lung cancer with either central (bronchogenic) or peripheral tumor location, and prior to surgery or other therapy for the cancer; Participants with a central or peripheral pulmonary recurrence of lung cancer following primary therapy may also be enrolled. Sputum samples for this cohort may be collected at or after a diagnostic bronchoscopy.

Exclusion Criteria:

* Severe obstructive lung disease
* Angina with minimal exertion
* Pregnancy
* Have or have had cancer other than lung cancer within one year
* Worked in the mining Industry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Dorian, BS Biology, Study Director; Lara Patriquin, MD, Principal Investigator — Radiology Associates of Albuquerquqe; Thomas Bauer, MD, Principal Investigator — Helen F Graham Cancer Center, Christiana Care
Locations (3):
- United States (3):
  - Waterbury Pulmonary Research, Waterbury, Connecticut
  - Helen F. Graham Cancer Center, Christiana Care Health System, Newark, Delaware
  - Radiology Associates of Albuquerque, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2009 to February 2011
  Helen F. Graham Cancer Center Newark, DE Christiana Care Health System, Newark, DE Waterbury Pulmonary Associates, Waterbury, CT
Groups:
- Single Arm Labeling of Deep-Lung Sputum Samples With TCPP: Deep-lung sputum was obtained from two cohorts, including (1) high-risk control group comprised of individuals not diagnosed but at high risk for lung cancer (n=102) and, (2) cancer group comprised of individuals with confirmed lung cancer diagnosis (n=26), was labeled in exact manner with TCPP and evaluated to detect red fluorescent [ie, cancer] cells (RFCs) from deep-lung sputum samples.
Period: Overall Study
Arm/Group | Single Arm Labeling of Deep-Lung Sputum Samples With TCPP
Started | 128
Completed | 128
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Male and female subjects aged 18 years of age and older were recruited from the pool of United States' military veterans who responded to public advertisements and recruitment pamphlets disseminated at veteran's events,
Arm/Group | Single Arm Labeling of Deep-Lung Sputum Samples With TCPP
Number analyzed (Participants) | 128
Age, Customized [Mean (Standard Deviation); unit: years]
  cohort 1 n=102 | 57.2 (11.6)
  cohort 2 n=26 | 61.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 111
Region of Enrollment [Number; unit: participants]
  United States | 128

OUTCOME MEASURES:

1. Primary Outcome: Determine the Clinical Sensitivity and Specificity of the Biomoda CyPath™ Early Lung Cancer Detection Assay Using Sputum Specimens From Two Cohorts of Participants and Estimate the Required Sample Size to Finalize a Protocol for a Pivotal Study.
Description: Various measurements were taken to report the validity of the findings. Sensitivity in this study was defined as the percentage of tumor cells that were positively identified. Specificity was the percentage of true positive signals and accuracy calculated as the percentage of those patients identified as having cancer.
  Testing for the study was performed at multiple locations to assess the efficacy of the CyPath Assay to detect lung cancer cells exfoliated from lung tumors present in deep-lung sputum. Participants who satisfied the inclusion/exclusion criteria were enrolled in the study and assigned to one of two cohorts (smoker with clear Low dose CT scan or "high-risk" normals," and lung cancer confirmed by pathology or "cancer").
Time Frame: March 2011
Measure: Number; unit: percentage
Groups:
- Single Arm Labeling of Deep-Lung Sputum Samples With TCPP: Deep-lung sputum was obtained from two cohorts, including (1) high-risk control group comprised of individuals not diagnosed but at high risk for lung cancer (n=102) and, (2) cancer group comprised of individuals with confirmed lung cancer diagnosis (n=26), was labeled in exact manner with TCPP and evaluated to detect red fluorescent [ie, cancer] cells (RFCs) from deep-lung sputum samples.
  CyPath: CyPath diagnostic assay for the early detection of lung cancer using sputum
Arm/Group | Single Arm Labeling of Deep-Lung Sputum Samples With TCPP
Number analyzed (Participants) | 128
percentage
  Sensitivity | 77.9
  Specificity | 65.7
  Accuracy | 81.3

ADVERSE EVENTS:
Arm/Group | Single Arm Labeling of Deep-Lung Sputum Samples With TCPP
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes